CLINICAL TRIAL: NCT05719506
Title: A Comparative Evaluation of Nebulized Dexmedetomidine and Nebulized Ketamine as a Premedication in Pediatric Surgeries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, alaa abohagar, Alaa Abo Hagar, M.D Lecturer of Anesthesia and Intensive Care,, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 34717/5/21
Record Dates: First submitted 2023-01-20; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Anesthesia Refusal
MeSH Terms: conditions — Treatment Refusal | interventions — Saline Solution; Pharmaceutical Preparations; Dexmedetomidine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group 1 (Sham Comparator): control group (nebulized normal saline without drug: group C) .The drugs will be prepared in 0.9% normal saline to a final volume of 3ml. Nebulization will be performed using a wall nebulizer and wall oxygen source on 4 l/min . A Research nurse who will not participate in the evaluation of sedation administered the drugs to all children in nebulizer sessions ∼30 min before transfer to the OR.
  Interventions: Other: normal saline without drug
- dexmedetomidine group 2 (Experimental): that receive nebulized dexmedetomidine (3 μg/kg; group D),The drugs will be prepared in 0.9% normal saline to a final volume of 3ml. Nebulization will be performed using a wall nebulizer and wall oxygen source on 4 l/min . A Research nurse who will not participate in the evaluation of sedation administered the drugs to all children in nebulizer sessions ∼30 min before transfer to the OR.
  Patients will be assessed for sedation score then separated from their parents and the ease of separation will be recorded.
  Interventions: Drug: Dexmedetomidine
- ketamine group 3 (Experimental): nebulized ketamine (3mg/kg; group K) ,The drugs will be prepared in 0.9% normal saline to a final volume of 3ml. Nebulization will be performed using a wall nebulizer and wall oxygen source on 4 l/min . A Research nurse who will not participate in the evaluation of sedation administered the drugs to all children in nebulizer sessions ∼30 min before transfer to the OR.
  Patients will be assessed for sedation score then separated from their parents and the ease of separation will be recorded.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Other: normal saline without drug — nebulizer session with normal saline only preoperative
  Other Names: control
  Arms: control group 1
Drug: Dexmedetomidine — nebulizer session with dexmedetomidine preoperative
  Other Names: precedex
  Arms: dexmedetomidine group 2
Drug: Ketamine — nebulizer session with ketamine preoperative
  Other Names: katalar
  Arms: ketamine group 3

SUMMARY:
preoperative anxiety and parental deprivation can be a traumatic time for young children undergoing surgery and remain challenges to anesthesiologists. Preoperative anxiety stimulates the sympathetic, parasympathetic, and endocrine systems, leading to an increase in heart rate (HR), blood pressure, and cardiac excitability. Pediatric anesthesiologists strive to minimize distress for children in the operating room (OR) environment and to provide a smooth induction of anesthesia

DETAILED DESCRIPTION:
This prospective double-blind randomized controlled study will be carried out in Tanta University Hospitals in Anesthesia Department from July 2021 to december 2021 on pediatric patients undergoing surgeries.

A written informed consent will be obtained from all patient parents who will receive an explanation to the purpose of the study and will have a secret code number to ensure privacy to participants and confidentiality of data.

Research results will be only used for scientific purposes. Procedures will be approved by both the Institutional and the Regional ethical committees.

Any unexpected risk appears during the course of the research will be cleared to the participants and ethical committee on time and proper measures will be taken to overcome or minimize these risks.

Randomization will be performed using the sealed opaque envelope technique; each patient's parent randomly selected a sealed envelope containing a group number in which the patient will be enrolled.

The sample size was calculated based on the following criteria:

* 95% confidence limit.
* 95% power of the study.
* The groups ratio is 1:1:1
* Based on a previous study , 18 patients in each group should be sufficient to detect a difference between means of the Ramsay sedation scale of 0.6 and a common standard deviation of 0.48.
* 2 cases were added to each group to overcome dropout. Therefore, we will recruit 20 cases in each group.

Anesthetic management: Preoperative assessment:

Which will include:

1. History :

   Clinical information such as age, gender, weight and other comorbidities will be evaluated.

   Take an 'AMPLE' history (allergies, medications, past medical/ anesthesia history, last meal, events leading up to the presentation), and ask about family history of problems with anesthesia.
2. Clinical examination Detailed airway assessment will be done.
3. Laboratory investigations Complete blood picture , bleeding time and clotting time . *All patients will be fasting for 2hr for clear fluids and 6-8 hr for solids.

Premedication:

In PACU, All the children will be monitored for heart rate, pulse oximetery and non-invasive blood pressure. All the baseline parameter will be observed and recorded.

Randomization:

Using sealed envelopes, patients will be assigned randomly to three groups (n=20 /group) that receive nebulized dexmedetomidine (3 μg/kg; group D) , nebulized ketamine (3mg/kg; group K) , control group (nebulized normal saline without drug: group C) .The drugs will be prepared in 0.9% normal saline to a final volume of 3ml. Nebulization will be performed using a wall nebulizer and wall oxygen source on 4 l/min . A Research nurse who will not participate in the evaluation of sedation administered the drugs to all children in nebulizer sessions ∼30 min before transfer to the OR.

Patients will be assessed for sedation score then separated from their parents and the ease of separation will be recorded.

In the OR:

Children will receive standard monitoring, including ECG, capnogram, noninvasive arterial blood pressure measurement and pulse oximetry.

Induction:

Induction of anesthesia will be done by inhalation of 8% sevoflurane in 100 % oxygen by anesthesia circuit, followed by the establishment of an intravenous peripheral line then i.v. fentanyl (1μg/kg) and atracurium (initial dose 0.5 mg/ kg) will be given and endotracheal tube will be inserted. Anesthesia will be maintained with 2% sevoflurane in a mixture of 50% air and 50% O2 to keep the end-tidal carbon dioxide pressure (PaCo2) between 30 and 35 mmHg and maintainence dose of atracurium (0.1 mg/ kg). When the surgery will end , sevoflurane discontinue, and residual neuromuscular blockade will be antagonized with IV atropine 0.02 mg/kg and IV prostigmine 0.05 mg/kg then tracheal extubation will be done and recovery time will be recorded. All patients will be transferred to PACU after tracheal extubation and discharge time will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* The children included in this study:

  * Will be of either gender.
  * Age between 3 and 10 years.
  * Belonging to American Society of Anesthesiologists (ASA) I, II physical status.
  * Undergoing elective surgery ranging in time between 30 - 90 minutes under general anesthesia.

Exclusion Criteria:

* Parental refusal of participation.
* Chest infection or respiratory distress.
* Cardiac disease.
* Mental or physical disability.
* Treatment with sedatives or anticonvulsants.
* Allergy to drugs or their ingredients.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
the sedating effects of these drugs . | 30 minutes
  the sedating effects of these drugs using Ramsay sedation scale as a premedications. Our target score (2 or 3 or 4) on the other side score 1 failure of sedation and score 5 or 6 over sedation.
  Table :Ramsay sedation scale
  1. Anxious and agitated, restless, or both.
  2. Cooperative, oriented, and calm.
  3. Responsive to commands only.
  4. Exhibiting brisk response to light glabellar tap or loud auditory stimulus.
  5. Exhibiting a sluggish response to light glabellar tap or loud auditory stimulus.
  6. Unresponsive.

SECONDARY OUTCOMES:
ease of parental separation | 30 minutes
  Patients also will be assessed for parental separation anxiety scale (PSAS) durig transferring the patient to OR. Score of 1 or 2 classified as an acceptable separation, whereas scores of 3 or 4 considered difficult separations from the parents.
  Table: Ease of parental separation and face mask Acceptance.
  1. Excellent: Patient unafraid, cooperative, or asleep
  2. Good :Slight fear and or crying, quiet with reassurance 3 -Fair :Moderate fear and crying, not quiet with reassurance
  4- Poor: Crying, need for restraint

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Tanta University Hospitals, Tanta
  - Tanta University, Tanta

IPD SHARING:
Plan to Share IPD: No
Once the study had been successfully completed, the data will be shared for other researchers.